CLINICAL TRIAL: NCT00400127
Title: The Effect of Silicone Suspension on Standing Balance for Transfemoral Amputees
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment, pilot outcome measures inappropriate
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: James Adderson, Capital District Health Authority, Canada
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CDHA015
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Amputee
Keywords: transfemoral amputee; silicon suspension; balance; gait

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- amputee (Experimental)
  Interventions: Device: Silesian suspension belt

INTERVENTIONS:
Device: Silesian suspension belt

SUMMARY:
The objective of this study is to test the hypothesis that silicone suction suspension without additional belt support does not significantly diminish the postural sway or walking performance of persons with transfemoral amputation.

ELIGIBILITY:
Inclusion Criteria:

* be forty-five (45) or older;
* unilateral transfemoral amputee;
* current patients of the QEII Health Sciences Centre Amputee Service based at the Rehab Site;
* can walk comfortably with their prosthesis for a minimum of 5 minutes, regardless of whether they require ambulation aids (i.e. canes, walkers, etc.);
* are in the process of being fitted with a silicon suction liner and pin system;
* are competent to give informed consent or have a proxy with power of attorney;
* have the written permission of the attending physician to participate;
* be willing to take part in the study, including signing the consent after carefully reading it.

Exclusion Criteria:

* have an unstable medical condition (e.g. angina, seizures), as determined by the attending or house physician;
* have major medical or neurological conditions that affect balance (specifically Parkinson's disease, stroke or Multiple Sclerosis), as determined by the physician or house staff physician;
* have an emotional or psychiatric problem of a type or extent that might make participation unpleasant, as determined by the attending or house physician.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Quiet standing balance
Timed-up and Go
ambulation profile
questionnaire

SECONDARY OUTCOMES:
demographics
prosthetic components

CONTACTS AND LOCATIONS:
Overall Officials: James Adderson, Principal Investigator — Capital Health, Canada
Locations (1):
- Nova Scotia Rehabilitation Centre, Halifax, Nova Scotia, Canada